CLINICAL TRIAL: NCT06487156
Title: FINN (First-line Ipilimumab + Nivolumab in NSCLC): An Italy, Nationwide, Prospective, Observational, Multicenter Study in Patients With First-line Nivolumab Plus Ipilimumab Therapy for Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate First-line Ipilimumab + Nivolumab in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Acronym: FINN
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-1409
Record Dates: First submitted 2024-06-06; First posted 2024-07-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Non-small cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants receiving first-line nivolumab plus ipilimumab
  Interventions: Drug: Nivolumab + ipilimumab

INTERVENTIONS:
Drug: Nivolumab + ipilimumab — As per product label

SUMMARY:
The purpose of this study is to collect and evaluate real-world data to describe the outcomes, patient characteristics, safety profile and treatment patterns of first-line nivolumab plus ipilimumab treatment for locally advanced or metastatic non-small cell lung cancer (NSCLC) in Italy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage IV or recurrent NSCLC (histologically or cytologically confirmed stage), without known EGFR- or ALK-alterations
* Decision to initiate a first-line treatment with nivolumab plus ipilimumab for the treatment of NSCLC according to the Italy label has been made independently of the study
* Patient is at least 18 years of age at time of treatment decision
* Patient provided written informed consent to participate in the study

Exclusion Criteria:

* Current primary diagnosis of a cancer other than NSCLC that requires systemic or other treatment
* Patients with known EGFR- or ALK-alterations
* Previous treatment with nivolumab and/or ipilimumab
* Patient already included in an interventional clinical trial for their advanced or recurrent NSCLC (but: Patients who have completed their participation in an interventional trial, who are not receiving study drug any more, and who are only followed-up for OS, can be enrolled)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with locally advanced or metastatic non-small cell lung cancer treated with nivolumab plus ipilimumab as first-line treatment
Sampling Method: Non-Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2030-10-11 (Estimated); Study Completion 2030-10-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 5 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 5 years
Overall response rate (ORR) | Up to 5 years
Best overall response (BOR) | Up to 5 years
Best overall response rate (BORR) | Up to 5 years
Tumor response to treatment as classified by the treating physician and Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Up to 5 years
Duration of response (DOR) | Up to 5 years
Time to response (TTR) | Up to 5 years
European Quality of Life-5 Dimensions (EQ-5D) Score | Baseline and up to 5 years
Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) results | Baseline and up to 5 years
Treatment regimen | Up to 5 years
Stage IV or recurrent, not previously treated, squamous and non-squamous NSCLC as confirmed by histology and/or cytology test results | Baseline
Number of participants discontinuing treatment | Up to 5 years
Management of Adverse Events (AEs) | Up to 5 years
Participant socio-demographic characteristics | Baseline and up to 5 years
Participant clinical characteristics | Baseline and up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts